CLINICAL TRIAL: NCT01980576
Title: Qualitative Pain Measurement and Sensitization at Patients With Degenerative Low Back Pain With Indication for Lumbar Intervertebral Disc
Brief Title: Qualitative Pain Measurement at Patients With Degenerative Low Back Pain
Status: Terminated | Type: Observational
Why Stopped: Lack of patients with the right criteria for inclusion
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: N-20110053
Record Dates: First submitted 2013-10-28; First posted 2013-11-11 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Degeneration of Lumbar Intervertebral Disc
Keywords: Pain; Sensitization; Spondylitis
MeSH Terms: conditions — Pain; Spondylitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pre-operative pain measurement: Patients with low back pain

SUMMARY:
The purpose of the study is:

* to measure sensitization of the nociceptive system at patients with low back pain in order to carry out a necessary surgical procedure
* to examine a possible association between low back pain and degenerative changes
* to analyse if low back pain is related to the clinical result 6 months after surgery
* to set up a model for pre-operative measurement of pain.

ELIGIBILITY:
Inclusion Criteria:

* patients who are going to be treated surgically for spondylitis
* ability to understand Danish in order to filling in a questionnaire
* a written signed statement of consent

Exclusion Criteria:

* removal of implants
* diabetic neuropathy or another neuropathic disease
* neurological diseases
* unability to read or understand Danish

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain measured at lumbar area, hip and ankle by an algometer | 6 months
  On basis of the extended examinations of low back pain, we expect to achieve a better knowledge to measure pain at this category of patients before a possible surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, M.D., Principal Investigator — Aalborg University Hospital, Denmark
Locations (1):
- Aalborg University Hospital, Aalborg, Region of Northern Jutland, Denmark